CLINICAL TRIAL: NCT04016116
Title: Study of PD-1 Inhibition With Pemrolizumab Alore or Combined With JAK 2 Inhibition in Myeloproliferative Neoplasm and Hodgkin's Lymphoma
Brief Title: Dual PD-1 and JAK2 Inhibition in Hematological Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01435
Record Dates: First submitted 2019-06-27; First posted 2019-07-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Cancer; Hematological Malignancy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — pembrolizumab; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab (Cohort 1) (Experimental): Pembrolizumab IV every 3 weeks (Cohort 1: Advanced progressive MPNs)
  Interventions: Drug: Pembrolizumab
- Pembrolizumab + Ruxolitinib (Experimental): Pembrolizumab IV every 3 weeks & Ruxolitinib po days 1-21 (Cohort 1: Advanced progressive MPNs)
  Interventions: Drug: Pembrolizumab; Drug: Ruxolitinib
- Pembrolizumab + Ruxolitinib (Cohort 2) (Experimental): Pembrolizumab IV every 3 weeks & Ruxolitinib po days 1-21 (Cohort 2, unresponsive to PD-1)
  Interventions: Drug: Pembrolizumab; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab IV every 3 weeks
  Other Names: keytruda
Drug: Ruxolitinib — Ruxolitinib po days 1-21
  Other Names: jakafi
  Arms: Pembrolizumab + Ruxolitinib; Pembrolizumab + Ruxolitinib (Cohort 2)

SUMMARY:
Pembrolizumab will have significant clinical activity in patients with Intermediate and high risk MF, advanced PV who have been resistant, failed or are intolerant to JAK2 inhibitor therapy and the activity may be enhanced in combination with JAK2 inhibition by Ruxolitinib; similarly MDS/MPN and CMML patients for who no standard therapies are available will exhibit responses to PD-1 or dual JAK2 and PD-1 treatment.

Adding JAK2 inhibitor Ruxolitinib to Pembrolizumab will have significant activity in patients with advanced, progressive HL who failed single agent PD-1 inhibition.

ELIGIBILITY:
Inclusion Criteria:

* advanced progressive MPNs, defined as intermediate and high risk MF or advanced PV resistant, failed or intolerant to JAK2 inhibitor therapy requiring medical therapy and patients with MDS/MPN Overlap and CMML having failed or for whom there are no standard therapies are available, are eligible. Patients will be allocated to one of two treatment arms:

  1. Pembrolizumab
  2. Pembrolizumab plus JAK2 inhibitor Ruxolitinib
* Patients with relapsed* or refractory* Hodgkin lymphoma (HL) who progress on PD-1 inhibitory treatment after achieving a partial response (PR) or complete response (CR) or stable disease (SD) or who are non-responsive to PD-1 inhibitory therapy. Patients must have failed appropriate standard treatment options.
* Relapsed: disease progression after most recent therapy
* Refractory: failure to achieve CR or PR to most recent therapy
* -The following laboratory values obtained less than 7 days prior to registration.

  * Total bilirubin ≤ 1.5 x Upper Limit normal (ULN) (except Gilbert's syndrome or known hemolysis or leukemic infiltration)
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN or < 5 x ULN if organ involvement
  * Alkaline Phosphatase < 5 x ULN
  * Serum creatinine ≤ 2 x ULN or 24 hour Cr clearance >60ml/min
  * Hematological inclusion criteria for:
  * MPN: -Platelet count ≥50,000/μL; Absolute neutrophil count (ANC) ≥250/μL
* Hematological inclusion criteria for:

  * MPN: -Platelet count ≥50,000/μL ;Absolute neutrophil count (ANC) ≥250/μL
  * MDS/MPN Overlap, CMML: Platelet count ≥25,000/μL; Absolute neutrophil count (ANC) ≥250/μ
  * HL-Platelet count ≥75,000/μL; Absolute neutrophil count (ANC) ≥1000/μL (800/ μL if marrow disease involvement; ECOG Performance Status (PS) 0 or 1 (Appendix I)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any of the following prior therapies:

  * Cytotoxic Chemotherapy less than 14 days prior to registration
  * Immunotherapy less than 14 days prior to registration
  * Biologic therapy (i.e. antibody therapies) less than 28 days prior to registration (see also 3.32)
  * Radiation therapy less than 14 days prior to registration
  * Targeted therapies (i.e. kinase inhibitors, less than 7 days or 5 half-life's whichever is shorter)
  * Hydroxyurea (HU) is allowed for blast count control throughout study
  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm ≤ 14 days prior to registration
* Active uncontrolled CNS leukemia. NOTE: Positive (cyto)pathology is allowed and patient can receive intrathecal chemotherapy
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy.
* Hypersensitivity to Ruxolitinib or any of its excipients.
* Acute Myeloid Leukemia with > 30% blasts in the bone marrow of peripheral blood
* Major surgery ≤ 28 days prior to treatment
* Clinically significant heart disease
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Pregnant women

* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Patients who have undergone an allogeneic stem cell transplantation within 5 years from registration are excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) measured using the Kaplan-Meier Method | 6 Months
  Progression free survival (PFS) is defined as the time from randomization or enrollment registration to the earliest date of documentation of disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Tibes, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States